CLINICAL TRIAL: NCT07061171
Title: The Impact of Continuous Positive Airway Pressure Combined With Physiotherapy on Ejection Fraction by Ameliorating Sleep Disturbance and Hypoxemia in Elderly Patients With Chronic Heart Failure and Obstructive Sleep Apnea: A Randomized Clinical Trial
Brief Title: CPAP and Physiotherapy for Heart Failure and Sleep Apnea in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weihua Peng (Other)
Responsible Party: Sponsor-Investigator, Weihua Peng, Principal investigator, Fugou County Minzhong Hospital
Organization: Fugou County Minzhong Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-B058
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Chronic Heart Failure; Obstructive Sleep Apnea
Keywords: Continuous Positive Airway Pressure; Physiotherapy; Elderly; Chronic Heart Failure; Obstructive Sleep Apnea; Sleep Disturbance
MeSH Terms: conditions — Sleep Apnea, Obstructive; Parasomnias | interventions — Continuous Positive Airway Pressure; Acupuncture Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group: CPAP plus Physiotherapy (Experimental): In addition to receiving the same CPAP therapy as the control group, patients in this arm received a 3-month physiotherapy regimen. The regimen consisted of: 1) Daily oral administration of a modified herbal decoction (Er Chen Tang with Chang Pu Yu Jin Tang); 2) Acupuncture sessions, once daily, 5 times per week; and 3) Head and occipital Tuina massage.
  Interventions: Device: Continuous Positive Airway Pressure; Drug: Herbal Decoction; Procedure: Acupuncture; Procedure: Tuina Massage
- Control Group: CPAP Alone (Active Comparator): Patients received CPAP therapy using a ResMed S9 AutoSet-S device. An optimal pressure or auto-adjusting range was determined via pressure titration. Patients were instructed to use the device for 5-7 hours per night, at least 5 nights per week, for 3 months. All patients also received standard conventional management for CHF and lifestyle advice.
  Interventions: Device: Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — Using a ResMed S9 AutoSet-S device with a pressure range of 4-20 cmH2O. Used for 5-7 hours per night, at least 5 nights per week, for 3 months.
Drug: Herbal Decoction — A daily dose of a decoction containing Ban Xia, Ju Hong, Shi Chang Pu, Yu Jin, Lai Fu Zi, Fu Ling, Bai Zhi, Cang Er Zi, and Gan Cao, administered orally in two divided doses.
  Arms: Study Group: CPAP plus Physiotherapy
Procedure: Acupuncture — Daily sessions with needle retention for 30 minutes, 5 times per week. Acupoints included Anmian (EX-HN22), Lianquan (CV23), Shanzhong (CV17), Zhongwan (CV12), Kongzui (LU6), Pishu (BL20), Fenglong (ST40), Zusanli (ST36), Yinlingquan (SP9), and Zhaohai (KI6).
  Arms: Study Group: CPAP plus Physiotherapy
Procedure: Tuina Massage — Includes massage techniques applied to the head and occipital region to relax muscles and improve local circulation.
  Arms: Study Group: CPAP plus Physiotherapy

SUMMARY:
This study evaluates whether adding physiotherapy (including herbal medicine, acupuncture, and Tuina massage) to standard continuous positive airway pressure (CPAP) therapy can provide superior benefits compared to CPAP alone for elderly patients suffering from both chronic heart failure (CHF) and obstructive sleep apnea (OSA). This randomized controlled trial aims to determine the combined therapy's efficacy and safety in improving sleep quality, hypoxemia, and cardiac function.

DETAILED DESCRIPTION:
The coexistence of chronic heart failure (CHF) and obstructive sleep apnea (OSA) in elderly patients creates a vicious cycle, worsening prognosis. Continuous positive airway pressure (CPAP) is the first-line treatment for OSA, but its efficacy in improving cardiac function in patients with comorbid CHF is debated. This prospective, randomized controlled trial was designed to evaluate the clinical efficacy of a comprehensive intervention combining CPAP with physiotherapy (herbal medicine, acupuncture, and Tuina massage). The study hypothesizes that this combined approach will be more effective than CPAP alone in improving sleep disturbances (assessed by the Pittsburgh Sleep Quality Index and Apnea-Hypopnea Index), alleviating hypoxemia (assessed by arterial blood gas analysis), and favorably modulating left ventricular ejection fraction (EF), thereby offering a superior management strategy for this complex patient population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CHF according to the New York Heart Association (NYHA) functional classification II-IV.
* Diagnosis of moderate to severe OSA (Apnea-Hypopnea Index [AHI] > 15 events/hour) confirmed by polysomnography.
* Age ≥ 65 years.
* Stable clinical condition for at least one month prior to enrollment.
* Ability to understand and comply with study procedures and provide informed consent.

Exclusion Criteria:

* Secondary hypertension.
* Acute myocardial infarction, congenital heart disease, rapid arrhythmias, significant valvular heart disease, cardiomyopathy, or severe hepatic/renal insufficiency.
* Other respiratory diseases such as chronic obstructive pulmonary disease (COPD), asthma, or pulmonary hypertension.
* Use of sedative drugs, morphine or its analogues, or other psychotropic medications; cognitive impairment.
* Received related treatment for OSA or significant changes in CHF medication within the past month.
* Withdrawal from the study midway.
* Current participation in other clinical drug trials.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 170 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Left Ventricular Ejection Fraction (EF) | Baseline and 3 months post-treatment
  Measured by echocardiography to compare the change in EF from baseline to 3 months post-treatment. EF (%) = (EDV - ESV) / EDV × 100%.
Change in Pittsburgh Sleep Quality Index (PSQI) Score | Baseline and 3 months post-treatment
  To assess sleep quality. The total score ranges from 0-21, with higher scores indicating poorer sleep quality.
Change in Apnea-Hypopnea Index (AHI) | Baseline and 3 months post-treatment
  Measured by overnight polysomnography, defined as the total number of apneas and hypopneas per hour of sleep.
Change in Arterial Oxygen Saturation (SaO2) | Baseline and 3 months post-treatment
  Measured via arterial blood gas analysis to assess improvement in hypoxemia.

SECONDARY OUTCOMES:
Change in End-Diastolic Volume (EDV) | Baseline and 3 months post-treatment
  Measured by echocardiography.
Change in End-Systolic Volume (ESV) | Baseline and 3 months post-treatment
  Measured by echocardiography.
Change in Epworth Sleepiness Scale (ESS) Score | Baseline and 3 months post-treatment
  To assess daytime sleepiness. The total score ranges from 0-24, with higher scores indicating greater sleepiness.
Change in Lowest Oxygen Saturation (LSaO2) | Baseline and 3 months post-treatment
  Measured by polysomnography.
Change in Longest Apnea Time (LAT) | Baseline and 3 months post-treatment
  Measured by polysomnography.
Change in Arterial Partial Pressure of Oxygen (PaO2) | Baseline and 3 months post-treatment
  Measured via arterial blood gas analysis.
Change in Arterial Partial Pressure of Carbon Dioxide (PaCO2) | Baseline and 3 months post-treatment
  Measured via arterial blood gas analysis.
Incidence of Adverse Reactions | During the 3-month treatment period
  Recording of all adverse events experienced during the treatment period, such as nasal itching, nasal dryness, dry eyes, or skin redness.

CONTACTS AND LOCATIONS:
Locations (1):
- Fugou County Minzhong Hospital, Zhoukou, Henan, China